CLINICAL TRIAL: NCT03575949
Title: Dual-Time Point (DTP) FDG PET CT for the Post-Treatment Assessment of Head and Neck Tumors Following Definitive Chemoradiation Therapy
Brief Title: Standard and Delayed FDG PET/CT After Chemoradiation Therapy in Assessing Patients With Metastatic Head and Neck Squamous Cell Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-0826; NCI-2018-02640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0826 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Malignant Neoplasm in the Spine
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (FDG PET/CT) (Experimental): Patients receive fludeoxyglucose F-18 IV over 1 minute and undergo PET/CT at 70 and 180 minutes after injection at 12-14 weeks following standard CRT completion.
  Interventions: Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo FDG PET/CT
  Other Names: CAT; CAT scan; Computerized Axial Tomography; computerized tomography; CT; CT scan; tomography
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well standard and delayed fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/computed tomography (CT) given after standard radiation and chemotherapy works in assessing patients with head and neck squamous cell cancer that has spread to other places in the body. Diagnostic procedures, such as PET/CT, use radioactive material, such as fludeoxyglucose F-18, to find and diagnose head and neck tumors and may help to find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the optimal imaging time using FDG positron emission tomography (PET) with comparison between a standard of care 1-hour scan (early) and the research scan of 3-hours scan (delayed) post radiotracer administration that maximizes separation of activity between lesion and non-lesional parenchyma (measured as lesion/background [L/B] ratio) in patients with head and neck primary squamous cell carcinoma following chemoradiation treatment.

OUTLINE:

Patients receive fludeoxyglucose F-18 intravenously (IV) over 1 minute and undergo PET/CT at 70 and 180 minutes after injection at 12-14 weeks following standard chemoradiation (CRT) completion.

After completion of study, patients are followed up at 30 days and then periodically for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult with computed tomography (CT) or fludeoxyglucose F-18 (FDG) positron emission tomography (PET) findings of cervical nodal metastasis from a head and neck primary squamous cell carcinoma treated with definitive chemoradiation

Exclusion Criteria:

* Children
* No evidence of cervical nodal metastasis
* Active infection of the head and neck
* Known allergy to FDG, iodine or gadolinium-based contrast agents
* Blood glucose (> 250 mg/dl)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Optimal imaging time | Up to 6 months
  Determined by fludeoxyglucose F-18 (FDG) positron emission tomography. The optimal time point is defined as the time point that meets the following requirements: 1) it has the largest average lesion/background (L/B) ratio, and 2) if the delayed time point is greater, it must be significantly different from the initial time point at the 0.025 significance level. The acquired PET data will be reconstructed using iterative techniques with resolution recovery. All delayed time points will then be registered using rigid techniques to the standard of care initial PET/CT image. Volumes of interest around the largest nodal metastasis will be drawn and the standard uptake value (SUV) max will be calculated. A corresponding region for largest nodal metastasis will be drawn on the contralateral sternocleidomastoid muscle respective to each lesion to determine L/B ratio, where L is the lesion SUV max and B is the corresponding background SUV max.
Differences in L/B ratio | Up to 6 months
  Differences in L/B ratio between the initial and delayed time point will be tested via paired t-test after appropriate transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Johnson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org